CLINICAL TRIAL: NCT03557138
Title: Study to Develop a Kinetic Model for FDG and Me4FDG in Kidneys of Type 2 Diabetic Patients With SGLT2 Inhibitor Therapies
Brief Title: Study to Develop a Kinetic Model for FDG and Me4FDG in Kidneys of Type 2 Diabetic Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. Marcus Hacker, Professor, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1128/2016
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Type2 Diabetes Mellitus
Keywords: SGLT2 inhibitor; 18F-FDG; alpha-Methyl-4-18F-FDG
MeSH Terms: interventions — methyl-4-fluoro-4-deoxyglucose

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Me4FDG (Experimental): Intravenous injection of alpha-Methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside (Me4FDG) and FDG for evaluation the kidney kinetic model of FDG and Me4FDG in type 2 diabetic patients with SGLT2-inhibitor therapies.
  Interventions: Behavioral: alpha-Methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside

INTERVENTIONS:
Behavioral: alpha-Methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside — positron emission tomography and magnetic resonance imaging (PET/MRI) of kidneys of diabetic patients using alpha-Methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside (Me4FDG)

SUMMARY:
In this study, using 18F-FDG and Gd-DTPA PET/MRI, we are aiming to perform a dynamic PET/MRI imaging using 18F-FDG and Me4FDG for a group of type 2 diabetic patients scheduled for Glifozine therapy due to the bad metabolic control to assess changes in renal function before and 1 to 2 weeks after initiating therapy with Gliflozine. Furthermore we aim to study the temporal behavior of 18F-FDG and Me4FDG activity in certain kidney regions of the diabetic participants to estimate basic kidney parameters using time activity curve. Further, we intend to find a kinetic model that describes the behavior of glucose in each part of the kidney can be acquired mathematically and to find out whether conclusions about the glucose reabsorption capability of the kidney in diabetes can be achieved in general. In addition, we aim to simultaneously determine renal lesions as well as obstructions with the fused, high definition, and three dimensional images of the kidney and estimate kidney function parameters from the dynamic Gd-DTPA MRI scan and compare them to the kidney function determined with the kinetic model.

DETAILED DESCRIPTION:
Independent of insulin, inhibition of sodium-glucose transporter 2 (SGLT2) in the proximal tubular cells prevents glucose reabsorption and promotes glucose excretion by causing glycosuria. Therefore, SGLT2 inhibitors known as Gliflozine are recently authorized for the treatment of type 2 diabetes mellitus (DM), whether as monotherapy or in combination with other anti-diabetic medications including insulin. To our knowledge, there is still no established kinetic model that describes precisely the reabsorption mechanism of glucose in the proximal tubules and that shows the impact of Gliflozine on renal function in diabetic patients. Therefore, the temporal behavior of glucose in the various kidney regions needs to be studied. Currently, the most promising tool is a combined positron emission tomography and magnetic resonance imaging (PET/MRI) using radioactive glucose analog 2-deoxy-2-(18F)fluoro-D-glucose (FDG). The MRI scan in combination with the kidney-specific gadolinium based contrast agent diethylenetriaminepentacetate (Gd-DTPA) images the organ with high resolution allowing an estimation of kidney parameters; the PET scan on the other hand shows the dynamic behavior of the glucose analog FDG. However, the reabsorption process of FDG in the kidney is controversial. For this reason, a dynamic PET/MRI image using 18F-FDG will be performed for diabetic patients, need the Gliflozine therapy, directly before and 1 to 2 weeks after therapy initiation. We aim, generally, to study the chronological behavior 18F-FDG activity in kidneys and to show, particularly, the reabsorption process under the influence of SGLT2 inhibition. Furthermore, conclusions about the glucose reabsorption capability of the kidney in these patients might be achieved and a kinetic model that describes the exact behavior of glucose in each part of the kidney can be mathematically acquired. We aim, additionally, to compare the PET/MRI images with the levels of diabetic metabolic control before and 1 to 2 weeks after initiating therapy with Gliflozine to show whether conclusions about therapy response can be drawn with FDG among the participants which arises from a broader peak in case of medication. A possible explanation is that the Patlak slope is among other influenced by the re-absorption process: if re-absorption is lowered due to the medication, the peak gets broader leading to a lower Patlak slope. We therefore conclude that reabsorption might be studied with FDG. Furthermore, a first draft of a kinetic model could be developed with the collected data According to this model, the re-absorption is mainly covered by the rate-constant k3. However, there was no correlation found between k3 and the above mentioned Patlak slope which most likely is a measure for re-absorption. Furthermore, the fit algorithm not always leads to meaningful results. This leads to the assumption that the model is not yet finished and further input data are needed. The model allows calculating the TACs of the visible renal sub-regions (Cortex, Medulla and Pelvis). In comparison with the measured TACs, the calculated ones deliver similar shapes. Although it seems from these results promising to study diabetes type II with a routine tracer like FDG, the kinetic model is hampered by the low affinity of FDG for the SGL transporter, which makes a quantification difficult. Therefore, an alternative radiopharmaceutical shall be applied which is similar to FDG but mainly re-abosrbed via SGLT: alpha-Methyl-4-[18F]FDG (Me4FDG).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM.
* Aged 20 -74 years.
* HbA1c level > 7%.
* Planned initiation of Gliflozine treatment.
* Intact renal function (serum creatinine < 1.5mg/dl or urinary albumin:creatinine ratio < 300mg/g in random urine sample).
* Written informed consent.

Exclusion Criteria:

* Age < 18 years, as kidneys may not be fully developed and not working properly yet.
* Impaired renal function (serum creatinine ≥ 1.5mg/dl or urinary albumin:creatinine ratio > 300mg/g in random urine sample) as well as anatomically altered or harmed kidneys could falsify the results due to their different or high alterable time activity curves.
* Patients under corticosteroids and diuretics therapies.
* MR-unsafe implants such as pacemakers and implantable cardioverter-defibrillators
* Intolerance of MRI contrast agents.
* Claustrophobia.
* Patients, who are not able to lie still without changing position for a minimum of 30 minutes.
* Pregnancy.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female diabetic patients with SGLT2-inhibitor therapies
Enrollment: 20 (Estimated)
Dates: Start 2017-02-22 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Kinetic behavior of glucose reabsorption | one year
  mathematically acquire a kinetic model of glucose reabsorption capability in each part of the kidney in type 2 diabetic patient under SGLT2-inhibitor therapies.

SECONDARY OUTCOMES:
positron emission tomography (PET) | one year
  Assess basic kidney parameters using time activity curve

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hacker, Prof., MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Radiology and Nuklear Medicine, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kobayashi M, Shikano N, Nishii R, Kiyono Y, Araki H, Nishi K, Oh M, Okudaira H, Ogura M, Yoshimoto M, Okazawa H, Fujibayashi Y, Kawai K. Comparison of the transcellular transport of FDG and D-glucose by the kidney epithelial cell line, LLC-PK1. Nucl Med Commun. 2010 Feb;31(2):141-6. doi: 10.1097/MNM.0b013e328333bcf5. PMID 19949354
- [Background] Geist BK, Baltzer P, Fueger B, Hamboeck M, Nakuz T, Papp L, Rasul S, Sundar LKS, Hacker M, Staudenherz A. Assessing the kidney function parameters glomerular filtration rate and effective renal plasma flow with dynamic FDG-PET/MRI in healthy subjects. EJNMMI Res. 2018 May 9;8(1):37. doi: 10.1186/s13550-018-0389-1. PMID 29744748
- [Derived] Geist BK, Ramirez JC, Binder P, Einspieler H, Ibeschitz H, Langsteger W, Nics L, Rausch I, Diemling M, Sohlberg A, Hacker M, Rasul S. In vivo assessment of safety, biodistribution, and radiation dosimetry of the [18F]Me4FDG PET-radiotracer in adults. EJNMMI Res. 2024 May 15;14(1):46. doi: 10.1186/s13550-024-01098-2. PMID 38750398
- [Derived] Rasul S, Geist BK, Brath H, Baltzer P, Sundar LKS, Pichler V, Mitterhauser M, Kautzky-Willer A, Hacker M. Response evaluation of SGLT2 inhibitor therapy in patients with type 2 diabetes mellitus using 18F-FDG PET/MRI. BMJ Open Diabetes Res Care. 2020 Mar;8(1):e001135. doi: 10.1136/bmjdrc-2019-001135. PMID 32205328